CLINICAL TRIAL: NCT06638346
Title: The Effect of Sex-specific Footwear and Tailored Injury Prevention Program on Cutting Performance
Brief Title: Effect of a Shortened FIFA11+ Warm-up Program and Sex-specific Footwear on Cutting in Youth Soccer Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: Natural Sciences and Engineering Research Council, Canada (Other); IDA sports (Unknown); Soccer Montréal (Unknown)
Responsible Party: Principal Investigator, Karen Chen, PhD Candidate, McGill University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: A12-M61-23B (23-10-088); RGPIN-2018-06525 (Other Grant/Funding Number: Natural Sciences and Engineering Research Council of Canada)
Record Dates: First submitted 2024-10-05; First posted 2024-10-15 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Healthy
Keywords: sidestep cutting; markerless motion capture system; injury prevention program; female-specific footwear; kinematics; shortened FIFA11+; youth soccer players

STUDY DESIGN:
Intervention Model Description: [Part1: Warm-up intervention]: It will consist of a longitudinal and prospective study conducted as a 2-group parallel quasi-randomized controlled trial with a 1:1 allocation and two time points (baseline, after 12-weeks). Both groups will complete a 12-week warm-up program. Group allocation will be done in a quasi-randomized fashion (see study detailed description).
  [Part2: Footwear study]: It will consist of a prospective, crossover design at one time point. All female participants will test both types of footwear (female-specific and unisex).
Masking Description: All the participants are within the same soccer organization and therefore complete masking of participants to group allocation is not possible. Coaches will be aware of allocations given that they will need to supervise the groups and give appropriate feedback if required. The primary investigator will be implicated in all aspects of the study (recruitment, data collection, supervision of training sessions, analysis) and thus will be aware of group allocations. Other research members that will help with data collection procedures will not be aware of group allocations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- [Part 1 of study]: Shortened FIFA 11+ Intervention Group (Experimental): The intervention group will complete a shortened FIFA11+ pre-activation training, incorporating 5 exercises from FIFA11+. The program will be performed twice a week for 12 weeks. The program lasts approximately 7 minutes.
  Interventions: Other: Shortened FIFA 11+ warm-up exercise program
- [Part 1 study]: Control Group (Standard warm-up) (Active Comparator): The control group will engage in a Brazilian warm-up, lasting approximately 7 minutes, 2 times a week for 3 months. Brazilian warm-ups are typically performed the usual warm-up routine at Soccer Montréal. A standardized version of the warm-up will be given so that all participants in the control group will undergo the same program.
  Interventions: Other: Brazilian warm-up exercise program

INTERVENTIONS:
Other: Shortened FIFA 11+ warm-up exercise program — The shortened FIFA11+ incorporates 5 exercises from the original FIFA11+ part 2 and 3: Sideways bench, single-leg stance, squats, jumping and plant and cut (refer to FIFA 11+ manual). All exercises, except plant and cut, have three levels of difficulty. Difficulty progression will follow FIFA11+ guideline option C where all players progress to the next level of all exercises after 3 or 4 weeks. This program is done on artificial turf.
  Coaches will be trained on FIFA guidelines by the primary investigator and provided with explanatory placards and the FIFA 11+ manual. The primary investigator will conduct checks twice a week with the coaches to address any questions and review the program. Only the shortened FIFA11+ group will receive verbal feedback as per FIFA11+ guidelines.
  Arms: [Part 1 of study]: Shortened FIFA 11+ Intervention Group
Other: Brazilian warm-up exercise program — The control group engages in a Brazilian warm-up. The warm-up consists of exercises performed in standing and while running including the following:
  * Performed in standing: Circular Arms (20-30 sec total), Opening and closing of the hips (20-30 sec total).
  * Performed while running back and forth on the field: Jogging (2 times), high kicks (2 times), glute kicks (2 times)
  * Performed while running forward (exercise), then small jog back without performing the exercise: hand-to-heel touches (2 times), knee and heel touches (2 times each side), side leg swings (2 times) and progressive sprint 80-90% speed (2 times).
  Coaches will supervise the session but will not be allowed to give verbal feedback. This program is done on artificial turf.
  Other Names: Usual soccer warm-up; Standard warm-up; Typical warm-up
  Arms: [Part 1 study]: Control Group (Standard warm-up)

SUMMARY:
This research aims to look at how warm-up programs and types of footwear affect movement patterns that are associated with injury risk during change-of-direction tasks, also known as cutting, in youth soccer players. Specifically, this research is conducted in two parts with two different study designs: a quasi-randomized controlled trial and a crossover design. The main questions it aims to answer are:

* [Part 1: Quasi-RCT] How does sex and a shortened FIFA11+ warm-up program, lasting 3 months, affect movement patterns during cutting compared to a standard warm-up program in youth soccer players?
* [Part 2: Crossover design] How does female-specific footwear affect movement patterns during cutting, compared to unisex footwear, in youth female players? Secondarily, whether specific shoe properties (comfort, functional traction, pressure distribution) differ between the two types of footwear.

For part 1 of the research:

* Researchers will compare a shortened FIFA11+ with a Brazilian warm-up program (standard) to see its effect on movement patterns during cutting.
* Participants will perform their assigned warm-up program twice a week for 3 months (12-weeks).
* To assess movement patterns, participants will perform an unplanned sidestep cutting task, captured with markerless cameras, before and after the training period.

For part 2, only female participants will be involved:

* Researchers will compare the effects of female-specific soccer cleats (designed exclusively for female) with unisex soccer cleats on cutting patterns and certain shoe properties.
* All participants will test both types of footwear and perform an unplanned sidestep task captured with markerless cameras, run through a slalom course (multiple acceleration and change of directions) to test for shoe traction, and complete an online survey on shoe comfort and perceived performance.
* A subset of participants will perform a planned sidestep task with wireless insoles to test for pressure distribution.

DETAILED DESCRIPTION:
With the rise of soccer's global prominence, injury risks among players remain a concern. Deceleration and change of direction maneuvers are frequently employed as an evasive strategy during games. However, they often contribute to higher risk of non-contact anterior cruciate ligament (ACL) injuries. Sidestep cutting involves planting with one foot and pushing off in the opposite direction. Improper movement patterns may increase loads on the planted leg leading to injuries. Injury prevention initiatives such as the FIFA11+ have been introduced to reduce injury rates, but it is unclear whether these programs can correct movement patterns during cutting. Moreover, the length of these programs (often lasting 20 minutes) can reduce adherence and hinder their practical implementation in the real-world. This results in alternative programs like the Brazilian warm-up to be used instead.

In addition, females are significantly more at-risk of ACL injuries than males. This is often attributed to differences in movement pattern and anatomy. Variations in foot anatomy can affect how players interact with footwear, which may in turn, influence cutting patterns. Yet, soccer footwear is typically designed using a male foot template (i.e. last), resulting in a one-size for all approach for female athletes.

In order to address current limitations, this study aims to estimate the effect of a shortened FIFA11+ and sex-specific footwear on cutting kinematics in youth soccer players. This will be done in two parts, where part 1 examines two warm-up programs, and part 2 examines two types of footwear. Ethics approval and informed participants and parental consent as well as assent have been obtained.

For part 1 of the study, 64 healthy soccer players will be recruited from Soccer Montréal (formerly known as Association Régionale de Soccer Concordia (ARSC)) sport study program. Soccer Montréal provides soccer sport study programs to high schools for high performance soccer players. Soccer Montréal conducts soccer training with pre-established cohorts separated by sex and age. Two male and 2 female cohorts will be allocated to either the intervention or control group. Male cohorts of similar age groups will be selected, and the entire cohort will be randomly allocated using a computer. The female cohorts have different age groups, and thus allocation to intervention or control will be divided within each cohort following a quasi-randomized fashion. During the testing, participants are required to perform an unanticipated sidestep maneuver at 45 (±10) degrees on artificial turf. Data will be collected with markerless motion capture systems. A total of 7 trials will be captured in each direction, only 5 out of 7 will be analyzed.

For part 2 of the study, female participants from part 1 (32 females) will test two types of footwear: Female-specific and unisex soccer cleats. Testing will be done at one time point. Female-specific cleats are provided from IDA sports, specifically the IDA centra FG/AG model. Unisex cleats are the Nike Tiempo Legend 10 Academy. Proper fit of shoe sizes will be examined manually by the research team prior to testing. Kinematic data will be collected using the same unanticipated sidestep task as part 1. Additional testing will include a slalom course to examine functional traction of the shoes. Participants will complete an online comfort survey, following the slalom course, once for each shoe. A subset of female participants will also complete a sidestep cutting task with wireless insoles to measure pressure data.

Findings of this study will advance knowledge of ACL injury mechanism during cutting tasks, aid in the design of more practical injury prevention programs and guide the development of female-specific footwear.

ELIGIBILITY:
Inclusion Criteria:

* Soccer players
* Enrolled in Association Régionale de Soccer Concordia (ARSC), now known as Soccer Montréal, soccer sport study program.
* Age between 13-17 years old.

Exclusion Criteria:

* Any history of major lower limb or back injuries (e.g., torn ACL, herniated vertebrae)
* History of any lower extremity surgery
* Current medical/neurological condition preventing cutting maneuver or training.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2024-01-29 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-05-22 (Actual)

PRIMARY OUTCOMES:
[Study Part 1: Warm-up programs]: Joint kinematics of lower extremity and trunk | At baseline
  Kinematic data will be captured for both intervention and control group using markerless motion capture system. Joint angles will be assessed throughout the cutting phase from pre-contact (100ms prior to foot strike) to foot-off of the planted leg. Specifically, joint kinematics will include: hip flexion/extension, hip abduction/adduction, hip internal/external rotation, knee flexion/extension, knee abduction/adduction, ankle dorsiflexion/plantarflexion, ankle inversion/eversion, trunk flexion/extension, trunk side flexion and trunk rotation.
  Principal component analysis will be used to analyze the whole angle waveform throughout cutting. Therefore, each kinematic outcome measure will be expressed as angle PC-scores which measures the degree of correspondence between angle waveform and principal components (PCs). PCs will captures variability features of angle waveform data such as amplitude, angle differences, etc.
[Study Part 1: Warm-up programs]: Joint kinematics of lower extremity and trunk | After the 12-week intervention
  Kinematic data will be captured for both intervention and control group using markerless motion capture system. Joint angles will be assessed throughout the cutting phase from pre-contact (100ms prior to foot strike) to foot-off of the planted leg. Specifically, joint kinematics will include: hip flexion/extension, hip abduction/adduction, hip internal/external rotation, knee flexion/extension, knee abduction/adduction, ankle dorsiflexion/plantarflexion, ankle inversion/eversion, trunk flexion/extension, trunk side flexion and trunk rotation.
  Principal component analysis will be used to analyze the whole angle waveform throughout cutting. Therefore, each kinematic outcome measure will be expressed as angle PC-scores which measures the degree of correspondence between angle waveform and principal components (PCs). PCs will captures variability features of angle waveform data such as amplitude, angle differences, etc.
[Study Part 2: Footwear]: Joint kinematics of lower extremity and trunk | Baseline (one time point)
  Kinematic data will be collected for female-specific footwear and unisex footwear using markerless motion capture system. Joint angles will be assessed throughout the cutting phase from pre-contact (100ms prior to foot strike) to foot-off of the planted leg. Specifically, joint kinematics will include: hip flexion/extension, hip abduction/adduction, hip internal/external rotation, knee flexion/extension, knee abduction/adduction, ankle dorsiflexion/plantarflexion, ankle inversion/eversion, trunk flexion/extension, trunk side flexion and trunk rotation.
  Principal component analysis will be used to analyze the whole angle waveform throughout cutting. Therefore, each kinematic outcome measure will be expressed as angle PC-scores which measures the degree of correspondence between angle waveform and principal components (PCs). PCs will capture variability features of angle waveform data such as amplitude, angle differences, etc.

SECONDARY OUTCOMES:
[Study Part 2: Footwear]: Slalom course running time | Baseline (one time point)
  Completion times will be captured with timing gates for both female-specific and unisex cleats. Faster completion times will reflect better functional traction properties. The average of three trials will be taken for each shoe.
[Study Part 2: Footwear]: Hindfoot mediolateral plantar pressure ratios | Baseline (one time point)
  Higher ratios will indicate greater relative pressure on the medial borders, while lower ratios will indicate greater pressures on the lateral border.
  Data will be determined for both for both female-specific and unisex cleats from the pressure data obtained with wireless insoles.
[Study Part 2: Footwear]: Forefoot mediolateral plantar pressure ratios | Baseline (one time point)
  Higher ratios will indicate greater relative pressure on the medial borders, while lower ratios will indicate greater pressures on the lateral border.
  Data will be determined for both for both female-specific and unisex cleats from the pressure data obtained with wireless insoles.
[Study Part 2: Footwear]: Peak plantar pressure | Baseline (one time point)
  The plantar surface of the foot will be divided into regions. Peak pressure will represent the highest recorded pressure in each of the regions.
  Data will be determined for both for both female-specific and unisex cleats from the pressure data obtained with wireless insoles.
[Study Part 2: Footwear]: Mean plantar pressure | Baseline (one time point)
  The plantar surface of the foot will be divided into regions. Mean pressure will be the average pressure in each of the regions.
  Data will be determined for both for both female-specific and unisex cleats from the pressure data obtained with wireless insoles.
[Study Part 2: Footwear]: Impulse plantar pressure | Baseline (one time point)
  Impulse (pressure-time integral) will be derived by multiplying the pressure amplitude by the duration of application (i.e. contact phase of interest).
  Data will be determined for both for both female-specific and unisex cleats from the pressure data obtained with wireless insoles.
[Study Part 2: Footwear]: Performance rating: Perceived traction suitability | Baseline (one time point)
  Perceived ratings will be completed using an online survey, following the slalom course, once for each shoe (female-specific and unisex cleats). Traction suitability rating ranges from 0 (Worse suitability) to 15 (Best suitability) using a visual analogue scale.
  Traction suitability refers to ability of the shoe to maintain its grip with the playing surface to minimize slip and falls. Worse suitability indicates greater slips and falls. Best suitability rating indicates a greater ability to maintain stability and less risk of slips and falls.
[Study Part 2: Footwear]: Performance rating: Overall performance | Baseline (one time point)
  Perceived ratings will be completed using an online survey, following the slalom course, once for each shoe (female-specific and unisex cleats). Overall performance rating ranges from 0 (Worse performance) to 15 (Best performance) using a visual analogue scale.
  Overall performance refers to how well you feel you did during the dynamic tasks in terms of overall speed, turn and satisfaction. Worse performance means that you did not perform well in this shoe. Best performance means that this shoe allowed you to give your best performance.
[Study Part 2: Footwear]: Comfort rating: Overall comfort | Baseline (one time point)
  Perceived ratings will be completed using an online survey, following the slalom course, once for each shoe (female-specific and unisex cleats). Overall comfort rating ranges from 0 (Not comfortable at all) to 15 (Most comfortable condition imaginable) using a visual analogue scale.
  Overall comfort refers to your overall impression of the shoe in terms of how comfortable. Not comfortable at all means that the shoe is overall not comfortable. Most comfortable condition imaginable, means that the shoe comfort is perfect for your needs.
[Study Part 2: Footwear]: Comfort rating: Overall shoe fit | Baseline (one time point)
  Perceived ratings will be completed using an online survey, following the slalom course, once for each shoe (female-specific and unisex cleats). Overall shoe fit rating ranges from 0 (Not comfortable at all) to 15 (Most comfortable condition imaginable) using a visual analogue scale.
  Shoe fit refers to the overall fit and size of the shoe. Not comfortable at all means the fit of the shoe is not comfortable either too tight or too loose at some parts of the foot. Most comfortable condition imaginable, means that the size and the fit of the shoe is perfect for your foot.
[Study Part 2: Footwear]: Comfort rating: Overall cushioning | Baseline (one time point)
  Perceived ratings will be completed using an online survey, following the slalom course, once for each shoe (female-specific and unisex cleats). Overall comfort rating ranges from 0 (Not comfortable at all) to 15 (Most comfortable condition imaginable) using a visual analogue scale.
  Overall cushioning refers to the softness/hardness of the insole at the forefoot or heel region. Not comfortable means the cushioning at the front or back of your foot is too hard or too soft, making it uncomfortable during use. Most comfortable means that the cushioning is perfectly fitted for your foot and needs.
[Study Part 2: Footwear]: Comfort rating: Overall shoe weight | Baseline (one time point)
  Perceived ratings will be completed using an online survey, following the slalom course, once for each shoe (female-specific and unisex cleats). Overall shoe weight rating ranges from 0 (Not comfortable at all) to 15 (Most comfortable condition imaginable) using a visual analogue scale.
  Shoe weight refers to the weight/heaviness of the shoe. Not comfortable at all means that the weight is too heavy or too light for your comfort. Most comfortable means that the shoe weight is perfect for your foot and tasks.

CONTACTS AND LOCATIONS:
Overall Officials: Shawn Robbins, Associate Professor, PhD, Study Director — McGill University; Karen Chen, PhD Candidate, Principal Investigator — McGill University
Locations (1):
- McGill University, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
The open-access content, encompass only de-identified biomechanical and demographic data. This will include metrics such as joint waveforms, plantar pressure, performance metrics, and anonymized demographic information including age, sex, height, weight, BMI, years of soccer experience, shoe size, and leg dominance.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Available following publication. No end date
Access Criteria: Our study data will be published in an open-access format (available to anyone who wishes to access the information), while protecting participant anonymity. It will encompass only de-identified biomechanical and demographic data, which will be shared via a dedicated repository on the McGill IHRG (Ice Hockey Research Group) server.

REFERENCES:
- [Background] Sterzing, T., Müller, C., Hennig, E. M., & Milani, T. L. (2009). Actual and perceived running performance in soccer shoes: A series of eight studies. Footwear Science, 1(1), 5-17. https://doi-org.proxy3.library.mcgill.ca/10.1080/19424280902915350
- [Background] Lam WK, Ng WX, Kong PW. Influence of shoe midsole hardness on plantar pressure distribution in four basketball-related movements. Res Sports Med. 2017 Jan-Mar;25(1):37-47. doi: 10.1080/15438627.2016.1258643. Epub 2016 Nov 21. PMID 27868427
- [Background] Kanko RM, Laende E, Selbie WS, Deluzio KJ. Inter-session repeatability of markerless motion capture gait kinematics. J Biomech. 2021 May 24;121:110422. doi: 10.1016/j.jbiomech.2021.110422. Epub 2021 Apr 8. PMID 33873117
- [Background] Ford, K. R., Nguyen, A. D., Westbrook, A. E., Mulrey, C. R., & Taylor, J. B. (2017). Footwear-induced changes in ankle biomechanics during unanticipated side-step cutting in female soccer players. Footwear Science, 9(sup1), S68-S70. https://doi-org.proxy3.library.mcgill.ca/10.1080/19424280.2017.1314343
- [Background] O'Brien J, Young W, Finch CF. The use and modification of injury prevention exercises by professional youth soccer teams. Scand J Med Sci Sports. 2017 Nov;27(11):1337-1346. doi: 10.1111/sms.12756. Epub 2016 Oct 7. PMID 27714907
- [Background] Soligard T, Nilstad A, Steffen K, Myklebust G, Holme I, Dvorak J, Bahr R, Andersen TE. Compliance with a comprehensive warm-up programme to prevent injuries in youth football. Br J Sports Med. 2010 Sep;44(11):787-93. doi: 10.1136/bjsm.2009.070672. Epub 2010 Jun 15. PMID 20551159
- [Background] Agel J, Rockwood T, Klossner D. Collegiate ACL Injury Rates Across 15 Sports: National Collegiate Athletic Association Injury Surveillance System Data Update (2004-2005 Through 2012-2013). Clin J Sport Med. 2016 Nov;26(6):518-523. doi: 10.1097/JSM.0000000000000290. PMID 27315457
- [Background] Carlson VR, Sheehan FT, Boden BP. Video Analysis of Anterior Cruciate Ligament (ACL) Injuries: A Systematic Review. JBJS Rev. 2016 Nov 29;4(11):e5. doi: 10.2106/JBJS.RVW.15.00116. PMID 27922985
- [Background] Wunderlich RE, Cavanagh PR. Gender differences in adult foot shape: implications for shoe design. Med Sci Sports Exerc. 2001 Apr;33(4):605-11. doi: 10.1097/00005768-200104000-00015. PMID 11283437
- See also: FIFA11+ Manual — https://kneesurgerysydney.com.au/wp-content/uploads/2017/05/11plus_workbook_e.pdf